CLINICAL TRIAL: NCT01529853
Title: Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Ascending Repeated Doses of SAR156597 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: To Evaluate the Effect of Different Doses of SAR156597 Given to Patients With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TDR11326; 2011-005481-37 (EudraCT Number); U1111-1124-1425 (Other: UTN)
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SAR156597 dose 1 (Experimental): SAR156597 dose 1, subcutaneous injection once every week
  Interventions: Drug: SAR156597
- SAR156597 dose 2 (Experimental): SAR156597 dose 2, subcutaneous injection once every week
  Interventions: Drug: SAR156597
- SAR156597 dose 3 (Experimental): SAR156597 dose 3, subcutaneous injection once every week
  Interventions: Drug: SAR156597
- Placebo (Placebo Comparator): Placebo (for SAR156597), subcutaneous injection once every week
  Interventions: Drug: Placebo (for SAR156597)

INTERVENTIONS:
Drug: SAR156597 — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: SAR156597 dose 1; SAR156597 dose 2; SAR156597 dose 3
Drug: Placebo (for SAR156597) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

To assess in adult patients with Idiopathic Pulmonary Fibrosis (IPF) the safety and tolerability of ascending doses of SAR156597 administered subcutaneously (SC) once weekly over a 6-week period.

Secondary Objectives:

To assess in adult patients with IPF:

* The pharmacodynamic effects of SAR156597, as measured on pulmonary function tests (PFTs), pulse oximetry and patient reported outcome and peripheral blood biomarkers.
* The trough plasma concentrations of SAR156597
* The potential immunogenicity of SAR156597.

DETAILED DESCRIPTION:
The study consists of a screening period of up to 28 days, treatment period of up to 6 weeks and a post-treatment follow-up period of up to 12 weeks. Total study duration is up to 22 weeks.

ELIGIBILITY:
Inclusion criteria:

* Adult (aged >18 years) male or female patients,
* Documented diagnosis of IPF according to the current American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/American Latin Thoracic Association (ATS/ERS/JRS/ALTA) guidelines

Exclusion criteria:

* Forced vital capacity (FVC) <50% of predicted value Carbon monoxide diffusing lung capacity (DLCO) (corrected for hemoglobin) <35% predicted value
* Oxygen saturation <90% by pulse oximetry while breathing ambient air at rest (sitting position for 10 min)
* Known diagnosis of significant respiratory disorders other than IPF
* Active vasculopathy or use of vasoactive drugs
* Known HIV or chronic viral hepatitis
* Patients with active tuberculosis or latent tuberculosis infection
* Evidence of any clinically significant, severe or unstable, acute or chronically progressive medical (other than IPF) or surgical disorder, or any condition that may affect patient safety in the judgment of the investigator
* Clinically significant abnormal ECG at screening
* Clinically significant laboratory tests at screening
* Current history of substance and/or alcohol abuse
* Females who are lactating or who are pregnant.
* Use of any registered therapy targeted to treat IPF within 4 weeks prior to screening
* Use of any cytotoxic/immunosuppressive agent including but not limited to azathioprine, cyclophosphamide, methotrexate and cyclosporine within 4 weeks prior to screening

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability: Number of participants with Adverse events | from first dose of study drug up to Week 18

SECONDARY OUTCOMES:
Pharmacodynamic: Change in forced (expiratory) vital capacity (FVC) | from baseline to week 6
Pharmacodynamic: Change in carbon monoxide diffusing lung capacity (DLco) | from baseline to week 6
Pharmacodynamic: Change in Saint George Respiratory Questionnaire (SGRQ) | from baseline to week 6
Pharmacodynamic: Change in plasma levels of biomarkers | from baseline to week 18
Pharmacokinetic: SAR156597 plasma concentration | from baseline to week 18

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (21):
- United States (11):
  - Investigational Site Number 840008, Sacramento, California
  - Investigational Site Number 840009, Jacksonville, Florida
  - Investigational Site Number 840011, Jacksonville, Florida
  - Investigational Site Number 840006, Chicago, Illinois
  - Investigational Site Number 840004, Joliet, Illinois
  - Investigational Site Number 840005, Maywood, Illinois
  - Investigational Site Number 840002, Wichita, Kansas
  - Investigational Site Number 840003, Minneapolis, Minnesota
  - Investigational Site Number 840013, New York, New York
  - Investigational Site Number 840014, Cincinnati, Ohio
  - Investigational Site Number 840010, Charleston, South Carolina
- Canada (3):
  - Investigational Site Number 124003, Edmonton
  - Investigational Site Number 124001, Hamilton
  - Investigational Site Number 124002, Vancouver
- Chile (3):
  - Investigational Site Number 152003, Santiago
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152002, Santiago
- Mexico (2):
  - Investigational Site Number 484003, Mexico City
  - Investigational Site Number 484002, Monterrey
- Spain (2):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724002, Barcelona